CLINICAL TRIAL: NCT04364113
Title: The Modification of Diet in Renal Disease Study
Acronym: MDRD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MDRD U01DK035073; U01DK035073 (NIH)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Chronic Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Study A Usual Protein Usual Pressure (Active Comparator): Study A Usual Protein and Usual Pressure
  Interventions: Other: Usual Protein Diet; Drug: Medications needed to maintain usual blood pressure
- Study A Usual Protein Low Pressure (Experimental): Study A Usual Protein and Low Pressure
  Interventions: Other: Usual Protein Diet; Drug: Medications needed to maintain low blood pressure
- Study A Low Protein Usual Pressure (Experimental): Study A Low Protein and Usual Pressure
  Interventions: Other: Low Protein Diet; Drug: Medications needed to maintain usual blood pressure
- Study A Low Protein Low Pressure (Experimental): Study A Low Protein and Low Pressure
  Interventions: Other: Low Protein Diet; Drug: Medications needed to maintain low blood pressure
- Study B Low Protein Usual Pressure (Active Comparator): Study B Low Protein and Usual Pressure
  Interventions: Other: Low Protein Diet; Drug: Medications needed to maintain usual blood pressure
- Study B Low Protein Low Pressure (Experimental): Study B Low Protein and Low Pressure
  Interventions: Other: Low Protein Diet; Drug: Medications needed to maintain low blood pressure
- Study B Very Low Protein Usual Pressure (Experimental): Study B Very Low Protein and Usual Pressure
  Interventions: Other: Very Low Protein Diet; Drug: Medications needed to maintain usual blood pressure
- Study B Very Low Protein Low Pressure (Experimental): Study B Very Low Protein and Low Pressure
  Interventions: Other: Very Low Protein Diet; Drug: Medications needed to maintain low blood pressure

INTERVENTIONS:
Other: Usual Protein Diet — The usual protein diet contains 1.30 g/kg/day protein and 16-20 mg/kg/day of Phosphorus
  Arms: Study A Usual Protein Low Pressure; Study A Usual Protein Usual Pressure
Other: Low Protein Diet — The low protein diet contains 0.575 g/kg/day protein and 5-10 mg/kg/day of Phosphorus
  Arms: Study A Low Protein Low Pressure; Study A Low Protein Usual Pressure; Study B Low Protein Low Pressure; Study B Low Protein Usual Pressure
Other: Very Low Protein Diet — The very low protein diet contains 0.28 g/kg/day or protein, mg/kg/day of Phosphorus and a keto acid mixture.
  Arms: Study B Very Low Protein Low Pressure; Study B Very Low Protein Usual Pressure
Drug: Medications needed to maintain usual blood pressure — The MAP goal for the usual blood pressure group is <=107 mm Hg for ages 18-60 and <=113 for ages 61+. Pharmacological and non-pharmacological therapies will be used to achieve the desired blood pressure values. The recommended anti-hypertensive regimen is a angiotensin-converting-enzyme inhibitor with or without a diuretic agent; a calcium-channel blocker or other medications can be added as needed.
  Arms: Study A Low Protein Usual Pressure; Study A Usual Protein Usual Pressure; Study B Low Protein Usual Pressure; Study B Very Low Protein Usual Pressure
Drug: Medications needed to maintain low blood pressure — The MAP goal for the low blood pressure group is <=92 mm Hg for ages 18-60 and <=98 for ages 61+. Pharmacological and non-pharmacological therapies will be used to achieve the desired blood pressure values. The recommended anti-hypertensive regimen is a angiotensin-converting-enzyme inhibitor with or without a diuretic agent; a calcium-channel blocker or other medications can be added as needed.
  Arms: Study A Low Protein Low Pressure; Study A Usual Protein Low Pressure; Study B Low Protein Low Pressure; Study B Very Low Protein Low Pressure

SUMMARY:
The Modification of Diet in Renal Disease Trial is a multicenter randomized clinical trial for men and women aged 18-70 years with chronic renal disease who are not on dialysis and who have not had a kidney transplant. Study participants are randomized in a 2 × 2 factorial design to diets containing different amounts of protein and phosphorus and to two levels of blood pressure control. The prescribed modifications differ depending on the level of a patient's kidney function. The primary outcome variable to compare diet or blood pressure groups is each patient's slope (or the change) in glomerular filtration rate (GFR) with time.

DETAILED DESCRIPTION:
Selection of patients is conducted in two periods: a screening period for initial determination of eligibility and a 3-month baseline period. The baseline period is used to instruct patients about study procedures; to assess GFR and dietary protein intake; and to control blood pressure according to standard medical practice. GFR, dietary protein, and urinary protein must meet the eligibility criteria at the end of the baseline period before an individual can be randomized.

Two different strata or studies are used depending on the level of an individual's GFR at the end of the baseline period. Study A is for individuals with a GFR from 25 to 55 ml/min/1.73 m^2 and a usual dietary protein intake of at least 0.90 g/kg/day, where kg are standard body weight. Study B is for persons with a baseline GFR from 13 to 24 ml/min/1.73 m^2 and no specification of protein intake.

Individuals who are randomized in the trial are prescribed one of three diets and one of two target mean arterial blood pressure goals (MAP). MAP is a weighted average of the diastolic and systolic blood pressures (two-thirds diastolic plus one-third systolic). The goals depend on the person's age. The moderate goal of 107 mm Hg is equivalent to a blood pressure of 140/90 mm Hg, the usual limits of normal blood pressure. The low-MAP goal of 92 mm Hg is a more strict level of control than usually achieved, equivalent to, for example, 125/75 mm Hg.

ELIGIBILITY:
Inclusion Criteria:

* Increased serum creatinine: Men: 1.4-7.0 mg/dl, Women: 1.2-7.0 mg/dl, or other objective evidence of kidney disease
* Mean arterial blood pressure <=125 mm Hg
* GFR 13-55 ml/min/1.73 m^2
* Urinary protein excretion <10 g/day
* Protein intake >0.90 g/kg/day if GFR 25-55 ml/min/1.73 m^2

Exclusion Criteria:

* Insulin-dependent diabetes or fasting serum glucose >200 mg/dl
* Patient on dialysis
* Kidney transplant recipient
* Lactating or pregnant woman or woman planning to become pregnant within the time frame of the study
* Doubtful compliance
* Body weight <80% or >160% of standard body weight
* Serum albumin <3.0 g/dl
* Selected renal disorders: Upper or lower urinary tract obstruction, Renal artery stenosis, Branched or staghorn calculi, Cystinuria
* Serious medical conditions: Malignancy (excluding skin cancer) within 1 year, Heart failure, New York Heart Association class 3 or 4, Lung disease, Liver disease, Gastrointestinal disease, Chronic systemic infections, including AIDS, Collagen vascular disease (other than rheumatoid arthritis), Frequent hospitalizations or disability
* Drugs: Immunosuppressive agents, Corticosteroids in excess of replacement dosage for 2 months per year or more, Gold or penicillamine within past month, Salicylates: more than 20 tablets per week, Other nonsteroidal antiinflammatory agents more than 3 times per week in past 2 months, Investigational drugs
* Allergy to iothalamate or iodine
* Inability or unwillingness to give consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 1989-01-01 (Actual); Primary Completion 1993-01-31 (Actual); Study Completion 2000-12-31 (Actual)

PRIMARY OUTCOMES:
Change in GFR slope | Up to 4 years
  Slopes will be calculated on the basis of the final baseline GFR and all follow-up values without adjustment for body surface area

SECONDARY OUTCOMES:
Dialysis or kidney transplantation | 3 years
  Time to first dialysis or kidney transplantation
Death from any cause | 3 years
  Time to death from any cause
Time to kidney failure | Up to 10 years
  The onset of kidney failure was ascertained from the US Renal Data System (USRDS) and included starting dialysis or undergoing kidney transplant
Time to kidney failure or death | Up to 10 years
  The onset of kidney failure was ascertained from the US Renal Data System (USRDS) and included starting dialysis or undergoing kidney transplant. Data for death were obtained from the National Death Index

CONTACTS AND LOCATIONS:
Overall Officials: Gerald J Beck, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: Yes
Data and samples are available at the National Institute of Diabetes Digestive and Kidney Diseases (NIDDK) Central Repository
Supporting Information: Study Protocol, CSR, Analytic Code
URL: https://repository.niddk.nih.gov/studies/mdrd/?query=mdrd

REFERENCES:
- [Result] Klahr S, Levey AS, Beck GJ, Caggiula AW, Hunsicker L, Kusek JW, Striker G. The effects of dietary protein restriction and blood-pressure control on the progression of chronic renal disease. Modification of Diet in Renal Disease Study Group. N Engl J Med. 1994 Mar 31;330(13):877-84. doi: 10.1056/NEJM199403313301301. PMID 8114857
- [Result] Levey AS, Greene T, Beck GJ, Caggiula AW, Kusek JW, Hunsicker LG, Klahr S. Dietary protein restriction and the progression of chronic renal disease: what have all of the results of the MDRD study shown? Modification of Diet in Renal Disease Study group. J Am Soc Nephrol. 1999 Nov;10(11):2426-39. doi: 10.1681/ASN.V10112426. PMID 10541304
- [Result] Sarnak MJ, Greene T, Wang X, Beck G, Kusek JW, Collins AJ, Levey AS. The effect of a lower target blood pressure on the progression of kidney disease: long-term follow-up of the modification of diet in renal disease study. Ann Intern Med. 2005 Mar 1;142(5):342-51. doi: 10.7326/0003-4819-142-5-200503010-00009. PMID 15738453
- [Result] Levey AS, Greene T, Sarnak MJ, Wang X, Beck GJ, Kusek JW, Collins AJ, Kopple JD. Effect of dietary protein restriction on the progression of kidney disease: long-term follow-up of the Modification of Diet in Renal Disease (MDRD) Study. Am J Kidney Dis. 2006 Dec;48(6):879-88. doi: 10.1053/j.ajkd.2006.08.023. PMID 17162142